CLINICAL TRIAL: NCT04408885
Title: Rehabilitation Treatment of Anterior Cruciate Ligament Rupture
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Horsens Hospital (Other); Central Jutland Regional Hospital (Other); Regionshospitalet Silkeborg (Other); Herning Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Other Study IDs: Danish EC: 1-10-72-25-20
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rehabilitation — Non-surgical interventions to patients with an Anterior cruciate ligament injury. Rehabilitation regime is the regime provided by the physician at the rehabilitation clinic.

SUMMARY:
The purpose with this present study is to investigate the effect og a non-surgical regime in patients with an Anterior Cruciate ligament injury.

The effect will be measured by patient reported outcome scores, level of function and how many of the patients are converting to operative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament injury where rehabilitation regime is selected as treatment.

Exclusion Criteria:

* Other knee ligament instability
* Rheumatoid arthritis
* Morbus Bechterews Disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will include 400 patients with Anterior cruciate ligament injury. Patients will be included at different orthopaedic Clinics at 5 hospitals in Region Midtjylland.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in patient reported outcome score (IKDC) | Baseline - 2 Years
  The International Knee Documentation Committee (0-100)

SECONDARY OUTCOMES:
Changes in patient reported outcome score (KOOS) | Baseline - 2 Years
  Knee injury and Osteoarthritis Outcome Score (0-100)
Changes in patient reported outcome score (KNEES-ACL) | Baseline - 2 Years
  Knee Numeric-Entity Evaluation Score (0-100)
Changes in patient reported outcome score (TEGNER) | Baseline - 2 Years
  Activity scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will not be available for other researchers